CLINICAL TRIAL: NCT02646020
Title: Aprepitant vs. Desloratadine in Non-small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors Related Pruritus: A Prospective, Randomized Control, Double-blinded, Phase II Clinical Trial
Brief Title: Aprepitant vs. Desloratadine in EGFR-TKIs Related Pruritus Treatment
Acronym: EGFR-TKIs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, M.D. Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAPE001
Record Dates: First submitted 2015-12-10; First posted 2016-01-05 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: pruritus; Non-small Cell Lung Cancer; Receptor, Epidermal Growth Factor; tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pruritus | interventions — Aprepitant; desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant and placebo (Experimental): aprepitant 125mg d1, 80mg d3 and d5, along with placebo 5mg d1-d28;
  Interventions: Drug: Aprepitant; Drug: Placebo of desloratadine
- desloratadine and placebo (Active Comparator): placebo 125mg d1, 80mg d3 and d5, along with desloratadine 5mg d1-d28
  Interventions: Drug: Desloratadine; Drug: Placebo of aprepitant

INTERVENTIONS:
Drug: Aprepitant — aprepitant 125mg d1, 80mg d3 and d5; until pruritus recurrence or discontinuation of EGFR-TKI or safely issues (SAE etc.)
  Other Names: Treatment arm: Aprepitant administration
  Arms: Aprepitant and placebo
Drug: Desloratadine — Desloratadine 5mg d1-d28; until pruritus recurrence or discontinuation of EGFR-TKI or safely issues (SAE etc.)
  Other Names: Treatment arm: Desloratadine administration
  Arms: desloratadine and placebo
Drug: Placebo of aprepitant — Placebo of aprepitant 125mg d1, 80mg d3 and d5; until pruritus recurrence or discontinuation of EGFR-TKI or safely issues (SAE etc.)
  Other Names: Comparative arm: Placebo of aprepitant administration
  Arms: desloratadine and placebo
Drug: Placebo of desloratadine — Placebo of desloratadine 5mg d1-d28; until pruritus recurrence or discontinuation of EGFR-TKI or safely issues (SAE etc.)
  Other Names: Comparative arm: Placebo of Desloratadine administration
  Arms: Aprepitant and placebo

SUMMARY:
Study hypothesis is that aprepitant is more effective than desloratadine in relieving pruritus caused by EGFR TKIs. Primary endpoint is the effective rate of pruritus, effective treatment defined as visual analogue scale (VAS) decrease ≥ 50% after treatment compared to baseline score. 130 NSCLC patients undertaken EGFR-TKI and suffer from moderate or severe pruritus (VAS score ≥ 4) will be enrolled in this study, and stratified (gender, VAS 4-6 or 7-10, and 2nd generation TKI or non 2nd generation) randomized (1:1) into aprepitant or desloratadine treatment. VAS investigation will be taken once a week to treatment end (4 weeks).

DETAILED DESCRIPTION:
This is a prospective, randomized control, double-blinded, phase II clinical trial. Study hypothesis is that aprepitant is more effective than desloratadine in relieving pruritus caused by EGFR TKIs. Primary endpoint is the effective rate of pruritus, effective treatment defined as visual analogue scale (VAS) decrease ≥ 50% after treatment (1 week) compared to baseline score. The VAS inquiry will be taken once a week for 4 weeks. Quality of life investigation will be performed at baseline, 1 week and 4 weeks after treatment using SKINDEX-16 questionnaire. 130 NSCLC patients undertaken EGFR-TKI and suffer from moderate or severe pruritus (VAS score ≥ 4) will be enrolled in this study, and stratified (gender,and VAS 4-6 or 7-10, and 2nd generation TKI or non 2nd generation) randomized (1:1) into aprepitant or desloratadine treatment. Aprepitant arm will be administrated aprepitant 125mg d1, 80mg d3 and d5, along with placebo 5mg d1-d28; desloratadine arm will be administrated placebo 125mg d1, 80mg d3 and d5, along with desloratadine 5mg d1-d28. Tolerance evaluation will be taken according to National Cancer Institute (NCI)-Common Terminology Criteria (CTC) For Adverse Events (AE) V4.03.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic non small cell lung cancer
* Undertaken EGFR TKIs treatment (gefitinib, erlotinib, icotinib, afatinib, etc)

  * 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Moderate or severe pruritus (VAS score ≥ 4) first occur after EGFR TKIs treatment
* Life expectancy ≥ 3 months
* Orally drug administration with no difficulty
* pregnancy test negative in 7 days for women of child-bearing age; willing to take contraception measures.
* Signed informed consent form (ICF)

Exclusion Criteria:

* Systemically treatment with Neurokinin-1 (NK-1) receptor inhibitors, antihistamines drugs, antibiotics, cortical hormone therapy, antiepileptic drugs, immunosuppressive agents or other drugs might affect treatment in 4 weeks; or locally used of these drug in 2 weeks.
* Existing skin lesions not EGFR TKIs related, such as skin infection, chronic dermatitis, Systemic Lupus Erythematosus (SLE), lymphoma or other diseases.
* Total bilirubin ≥ 1.5 Upper Limit Of Normal (ULN)
* Serum creatinine ≥mg/dl
* AST or ALT ≥ 2.5 ULN without liver metastasis; or ≥ 5 ULN with liver metastasis.
* Residual toxicity event ≥ CTC-AE grade 2, except peripheral neurotoxicities.
* Central nervous system (CNS) metastasis or spinal compression; except no symptoms and with no cortical hormonotherapy in 4 weeks.
* Clinical evidence of interstitial lung disease
* Any severe or uncontrolled systemic diseases judged by investigators.
* Any contraindication of Neurokinin-1 receptor inhibitors and desloratadine.

Discontinuation Criteria

* Invalid subject after randomization
* Major protocol violations judged by investigators.
* Poor compliance
* Intolerable adverse events
* Subject withdraw ICF
* Any pregnancy events
* No clinical benefits due to clinical adverse events, laboratory abnormalities or other medical conditions
* Other reasons of treatment discontinuation judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-12; Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
effective rate of pruritus relieving | day 28 at the treatment ends
  effective treatment of pruritus relieving defined as visual analogue scale (VAS) decrease ≥ 50% after treatment compared to baseline score

SECONDARY OUTCOMES:
duration of pruritus relieving | 12 weeks at the follow-up end
  the time from pruritus effective relief to VAS score increase ≥ baseline level, the VAS inquiry will be taken once a week.
Change from baseline quality of life assessment at treatment ends | baseline, 28 days at the treatment ends
  using SKINDEX-16 questionnaire to assess patients quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Result] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Result] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Result] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771
- [Result] Zhang L, Ma S, Song X, Han B, Cheng Y, Huang C, Yang S, Liu X, Liu Y, Lu S, Wang J, Zhang S, Zhou C, Zhang X, Hayashi N, Wang M; INFORM investigators. Gefitinib versus placebo as maintenance therapy in patients with locally advanced or metastatic non-small-cell lung cancer (INFORM; C-TONG 0804): a multicentre, double-blind randomised phase 3 trial. Lancet Oncol. 2012 May;13(5):466-75. doi: 10.1016/S1470-2045(12)70117-1. Epub 2012 Apr 17. PMID 22512843
- [Result] Lynch TJ Jr, Kim ES, Eaby B, Garey J, West DP, Lacouture ME. Epidermal growth factor receptor inhibitor-associated cutaneous toxicities: an evolving paradigm in clinical management. Oncologist. 2007 May;12(5):610-21. doi: 10.1634/theoncologist.12-5-610. PMID 17522250
- [Result] Lacouture ME, Anadkat MJ, Bensadoun RJ, Bryce J, Chan A, Epstein JB, Eaby-Sandy B, Murphy BA; MASCC Skin Toxicity Study Group. Clinical practice guidelines for the prevention and treatment of EGFR inhibitor-associated dermatologic toxicities. Support Care Cancer. 2011 Aug;19(8):1079-95. doi: 10.1007/s00520-011-1197-6. Epub 2011 Jun 1. PMID 21630130
- [Result] Chan A, Tan EH. How well does the MESTT correlate with CTCAE scale for the grading of dermatological toxicities associated with oral tyrosine kinase inhibitors? Support Care Cancer. 2011 Oct;19(10):1667-74. doi: 10.1007/s00520-010-0999-2. Epub 2010 Sep 5. PMID 20820812
- [Result] Ocvirk J, Cencelj S. Management of cutaneous side-effects of cetuximab therapy in patients with metastatic colorectal cancer. J Eur Acad Dermatol Venereol. 2010 Apr;24(4):453-9. doi: 10.1111/j.1468-3083.2009.03446.x. Epub 2009 Sep 27. PMID 19793151
- [Result] Scope A, Agero AL, Dusza SW, Myskowski PL, Lieb JA, Saltz L, Kemeny NE, Halpern AC. Randomized double-blind trial of prophylactic oral minocycline and topical tazarotene for cetuximab-associated acne-like eruption. J Clin Oncol. 2007 Dec 1;25(34):5390-6. doi: 10.1200/JCO.2007.12.6987. PMID 18048820
- [Result] Porzio G, Aielli F, Verna L, Porto C, Tudini M, Cannita K, Ficorella C. Efficacy of pregabalin in the management of cetuximab-related itch. J Pain Symptom Manage. 2006 Nov;32(5):397-8. doi: 10.1016/j.jpainsymman.2006.07.006. No abstract available. PMID 17085262
- [Result] Stander S, Siepmann D, Herrgott I, Sunderkotter C, Luger TA. Targeting the neurokinin receptor 1 with aprepitant: a novel antipruritic strategy. PLoS One. 2010 Jun 4;5(6):e10968. doi: 10.1371/journal.pone.0010968. PMID 20532044
- [Result] Stander S, Weisshaar E. Medical treatment of pruritus. Expert Opin Emerg Drugs. 2012 Sep;17(3):335-45. doi: 10.1517/14728214.2012.711316. Epub 2012 Aug 7. PMID 22870909
- [Result] Chang SE, Han SS, Jung HJ, Choi JH. Neuropeptides and their receptors in psoriatic skin in relation to pruritus. Br J Dermatol. 2007 Jun;156(6):1272-7. doi: 10.1111/j.1365-2133.2007.07935.x. PMID 17535226
- [Result] Quartara L, Altamura M. Tachykinin receptors antagonists: from research to clinic. Curr Drug Targets. 2006 Aug;7(8):975-92. doi: 10.2174/138945006778019381. PMID 16918326
- [Result] Booken N, Heck M, Nicolay JP, Klemke CD, Goerdt S, Utikal J. Oral aprepitant in the therapy of refractory pruritus in erythrodermic cutaneous T-cell lymphoma. Br J Dermatol. 2011 Mar;164(3):665-7. doi: 10.1111/j.1365-2133.2010.10108.x. Epub 2011 Jan 28. No abstract available. PMID 21039410
- [Result] Vincenzi B, Fratto ME, Santini D, Tonini G. Aprepitant against pruritus in patients with solid tumours. Support Care Cancer. 2010 Sep;18(9):1229-30. doi: 10.1007/s00520-010-0895-9. Epub 2010 Jun 11. No abstract available. PMID 20544226
- [Result] Jimenez Gallo D, Albarran Planelles C, Linares Barrios M, Fernandez Anguita MJ, Marquez Enriquez J, Rodriguez Mateos ME. Treatment of pruritus in early-stage hypopigmented mycosis fungoides with aprepitant. Dermatol Ther. 2014 May-Jun;27(3):178-82. doi: 10.1111/dth.12113. Epub 2013 Dec 2. PMID 24517320
- [Result] Santini D, Vincenzi B, Guida FM, Imperatori M, Schiavon G, Venditti O, Frezza AM, Berti P, Tonini G. Aprepitant for management of severe pruritus related to biological cancer treatments: a pilot study. Lancet Oncol. 2012 Oct;13(10):1020-4. doi: 10.1016/S1470-2045(12)70373-X. Epub 2012 Sep 18. PMID 22995650
- [Result] Marquez D, Ramonda C, Lauxmann JE, Romero CA, Vukelic VL, Martinatto C, Barron B, Novoa PA, Peixoto AJ, Orias M. Uremic pruritus in hemodialysis patients: treatment with desloratidine versus gabapentin. J Bras Nefrol. 2012 Jun;34(2):148-52. doi: 10.1590/s0101-28002012000200007. PMID 22850916
- [Result] Bachert C, Maurer M. Safety and efficacy of desloratadine in subjects with seasonal allergic rhinitis or chronic urticaria: results of four postmarketing surveillance studies. Clin Drug Investig. 2010;30(2):109-22. doi: 10.2165/11530930-000000000-00000. PMID 20067329
- [Result] Grob JJ, Auquier P, Dreyfus I, Ortonne JP. Quality of life in adults with chronic idiopathic urticaria receiving desloratadine: a randomized, double-blind, multicentre, placebo-controlled study. J Eur Acad Dermatol Venereol. 2008 Jan;22(1):87-93. doi: 10.1111/j.1468-3083.2007.02385.x. PMID 18181978
- [Result] Ortonne JP, Grob JJ, Auquier P, Dreyfus I. Efficacy and safety of desloratadine in adults with chronic idiopathic urticaria: a randomized, double-blind, placebo-controlled, multicenter trial. Am J Clin Dermatol. 2007;8(1):37-42. doi: 10.2165/00128071-200708010-00005. PMID 17298105
- [Derived] Zhou T, Zhang Y, Ma Y, Ma W, Wu X, Huang L, Feng W, Zhou H, Liu J, Zhao H, Zhang L, Yang Y, Huang Y. Comparison of aprepitant versus desloratadine for EGFR-TKI-induced pruritus: A randomized phase 2 clinical trial. Cancer. 2022 Nov 15;128(22):3969-3976. doi: 10.1002/cncr.34474. Epub 2022 Oct 5. PMID 36197287